CLINICAL TRIAL: NCT06739629
Title: The School Meal Intervention: the Effect of Yellow Mealworm-enriched Maize Porridge on Nutrition and Health Status of 6-9-year-old Children
Brief Title: Refugee Insect Production for Food and Feed: the School Meal Intervention
Acronym: REFIPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Makerere University (Other); International Centre of Insect Physiology and Ecology (ICIPE) (Other); Mothers Against Malnutrition and Hunger (Unknown); Child and Family Health, Uganda (Unknown); Research and Action for Income Security (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: S400- REFIPRO STUDY
Record Dates: First submitted 2024-11-22; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: Two-arm randomized intervention
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Data collectors assessing anthropometric measures, dietary records and questionnaires were masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yellow mealworm-enriched porridge (Experimental): Participants receive a daily meal of yellow mealworm-enriched porridge, served in schools. The porridge provides 420 Kcal/serving
  Interventions: Other: Insect porridge
- Maize porridge (Other): Participants receive a standard maize porridge served in schools. This porridge is comparable to the porridge served in the parent-led school feeding program.
  Interventions: Other: Maize Porridge

INTERVENTIONS:
Other: Insect porridge — Yellow mealworm porridge
  Other Names: Yellow mealworm porridge; Edible insect porridge
  Arms: Yellow mealworm-enriched porridge
Other: Maize Porridge — Maize porridge
  Other Names: porridge
  Arms: Maize porridge

SUMMARY:
The goal of this randomized controlled trial is to assess whether edible insect-enriched school porridge has nutrition and health benefits for children aged 6-9 years in refugee communities in Uganda.

The main question the research aims to answer is: Does a daily serving of maize porridge enriched with yellow mealworm flour improve the gut health, growth, and micronutrient status of children in comparison to a standard maize porridge?

Participants will:

Consume a daily serving of yellow mealworm porridge or a maize porridge for one school term (3 months). Data is collected before, during and after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Children in Primary 1 in Bukere and Kako primary school
* Age: 6-9 years
* Child can eat insects
* Written informed consent given by parent/caregiver

Exclusion Criteria:

* Severe acute malnutrition measured as MUAC < 13.5 cm
* Known allergies related to consuming insects
* Disability that impedes eating capacity
* Disability that makes height assessment problematic
* Family plans to move away or deregister child from Kako and Bukere primary schools within the school term.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in linear growth based on absolute height gain over 3 months intervention period | 3 months
  Assessing the effect of the intervention on height gain measured in cm

SECONDARY OUTCOMES:
Change in myeloperoxidase (MPO) over 3 months intervention period | 3 months
  Assessing the effect of the intervention on myeloperoxidase (ng/mL), which is a stool marker for Environmental Enteric Dysfunction (EED). A high value indicates high intestinal inflammation.
Change in alpha-1-anti-trypsin (AAT) over 3 months intervention period | 3 months
  Assessing the effect of the intervention on alpha-1-anti-trypsin (mg/g) which is a stool marker for Enteric Environemtal Dysfunction ( EED). A high value indicates high intestinal protein loss.
Change in in Neopterin (NEO) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on Neopterin ( nmol/L) which is a stool marker for Enteric Environemtal Dysfunction (EED). A high value indicates intestinal inflammation.
Change in weight over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on weight gain (kg)
Change in BMI- for- age Z-score over 3 months intervention period | 3 months
  Assessing the effect of the intervention on BMI-for-age Z-score, by combining weight (Kg) and Height (m2) to report BMI (kg/m2) using the cut offs: Overweight: >+1SD, Obesity: >+2SD, Thinness: <-2SD, Severe thinness: <-3SD
Change in Height- for-age Z-score over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on height-for-age Z-score values using the cut offs: < -2 to -3 HAZ moderately stunted, HAZ < -3 severely stunted
Change in Weight- for-age Z-score over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on weight-for-age Z-score using the cut offs: -2 to-3 WAZ moderately underweight, WAZ < -3 severely underweight
Change in Mid-Upper Arm Circumference (MUAC) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on the Mid-Upper Arm Circumference in cm using the cut-offs: <13.5cm severe acute malnutrition, 13.5cm -14.5cm moderate acute malnutrition.
Change in Subscapular and Triceps skinfold thickness over 3 months intervention period | 3 months
  Assessing the effect of the intervention on subscapular and triceps skinfold thickness measured in mm.
Change in waist circumference measurement over 3 months intervention period | 3 months
  Assessing the effect of the intervention on waist circumference measured in cm.
Change in fat mass over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on fat mass measured in kgs using deuterium dilution method and bioimpedance analyzer. Low fat mass indicates healthier body composition.
Change in fat free mass over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on fat free mass measured in kg using deuterium dilution method and bioimpedance analyzer. A high fat free mass indicates high muscle mass and healthier body composition.
Change in fat mass index over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on fat mass index measured in kg/m2, using deuterium dilution method and bioimpedance analyzer. Low fat mass index indicates a healthier body composition.
Change in fat free mass index over 3 months intervention period | 3 months
  Assessing the effect of the intervention on fat free mass index ( FFMI) measured in kg/m2 using deuterium dilution method and bioimpedance analyzer. A high fat free mass index indicates high muscle mass and healthier body composition
Change in C- reactive protein (CRP) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on C-reactive Protein(mg/L) which is a blood marker for systemic inflammation. High CRP values indicate systemic inflammation.
Change in alpha-1-acid glycoprotein (AGP) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on alpha-1-acid glycoprotein (g/L) which is a blood marker for systemic inflammation. High AGP values indicate systemic inflammation.
Change in insulin like growth factor (IGF-1) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on insulin like growth factor (ng/mL) which is a blood markers for growth. High IGF-1 values support growth.
Change in hemoglobin over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on hemoglobin measured in g/dL. Low hemoglobin levels indicate Anemia.
Change in ferritin over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on serum ferritin measured in μg/L. A low level of serum ferritin indicates Anemia.
Change in soluble transferrin receptor (sTfR) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on soluble transferrin receptor measured in mg/L. A high level of sTfR is associated with Anemia.
Change in cobalamin over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on cobalamin measured in pmol/L. A low level of cobalamin is associated with Vitamin B12 deficiency.
Change in retinol binding protein (RBP) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on serum retinol binding protein (RBP) measured in µmol/l. A low level of RBP is associated with Vitamin A deficiency.
Change in methyl malonic acid (MMA) over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on methyl malonic acid (MMA) measured in nmol/L. A high level of MMA indicates Vitamin B12 deficiency.
Change in citrulline over the 3 months intervention period | 3 months
  Assessing the effect of the intervention on plasma citrulline measured in μmol/L. A low level of citrulline indicates impaired intestinal function.

CONTACTS AND LOCATIONS:
Overall Officials: Ezekiel Mupere, PhD, MD, Principal Investigator — Makerere University
Locations (1):
- Kako and Bukere Primary School, Kyegegwa, Uganda

IPD SHARING:
Plan to Share IPD: No